CLINICAL TRIAL: NCT05771259
Title: Ody Contouring After Bariatric Surgeries in Jordan: Awareness, Prevalence, and Challenges
Brief Title: Body Contouring After Bariatric Surgeries in Jordan
Status: Completed | Type: Observational
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Amani Atallah, M.D, University of Jordan
Other Study IDs: 10/2023/5723
Record Dates: First submitted 2023-03-04; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Body Contouring

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Participants who didn't undergo body contouring surgery after bariatric surgery.
  Interventions: Other: Assessment of knowledge and behaviour
- Group B: Participants who underwent body contouring surgery after bariatric surgery.
  Interventions: Other: Assessment of knowledge and behaviour

INTERVENTIONS:
Other: Assessment of knowledge and behaviour — Assessment of knowledge and behaviour

SUMMARY:
This study aimed to describe Jordanians' awareness and knowledge of body-contouring surgeries and estimate their prevalence. Additionally, we aimed to identify the limitations reported by our population and compare them with those reported in the literature.

DETAILED DESCRIPTION:
We aimed to reach out to 351 patients who underwent bariatric surgery at JUH as well as an additional 100 patients who underwent BS at one of the largest private medical facilities in Amman between January and June of 2021. We distributed a validated questionnaire to all patients. Of the 451 patients, 305 completed the questionnaire (response rate: 67.6%). The inclusion criteria were age 13-63 years, BS type (sleeve gastrectomy or Roux-en-Y bypass), and completion of the questionnaire. Responses that did not meet these criteria or contained duplicates were excluded (n=11). The remaining 294 responses were collected and entered into a database for the analysis.Three main variables were assessed in each group in addition to multiple other observations. The main variables were sex, marital status, and employment status.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-63 years
* Bariatric surgery type (LSG or RYGB)

Exclusion Criteria:

* Incomplete or duplicate reponses
* Bariatric surgery ype (Gastric band)

Ages: 13 Years to 63 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Of the 451 patients, 305 completed the questionnaire (response rate: 67.6%). The inclusion criteria were age 13-63 years, BS type (sleeve gastrectomy or Roux-en-Y bypass), and completion of the questionnaire.
Sampling Method: Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Prevalence of Body contouring surgeries after bariatric surgeries | 07/2017-06/2021

CONTACTS AND LOCATIONS:
Locations (1):
- University of Jordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nguyen NT, Root J, Zainabadi K, Sabio A, Chalifoux S, Stevens CM, Mavandadi S, Longoria M, Wilson SE. Accelerated growth of bariatric surgery with the introduction of minimally invasive surgery. Arch Surg. 2005 Dec;140(12):1198-202; discussion 1203. doi: 10.1001/archsurg.140.12.1198. PMID 16365242
- [Background] Ellison JM, Steffen KJ, Sarwer DB. Body Contouring After Bariatric Surgery. Eur Eat Disord Rev. 2015 Nov;23(6):479-87. doi: 10.1002/erv.2408. Epub 2015 Sep 22. PMID 26395601
- [Background] Monpellier VM, Antoniou EE, Mulkens S, Janssen IMC, Jansen ATM, Mink van der Molen AB. Body Contouring Surgery after Massive Weight Loss: Excess Skin, Body Satisfaction, and Qualification for Reimbursement in a Dutch Post-Bariatric Surgery Population. Plast Reconstr Surg. 2019 May;143(5):1353-1360. doi: 10.1097/PRS.0000000000005525. PMID 30789477
- [Background] Derderian SC, Patten L, Kaizer AM, Inge TH, Jenkins TM, Michalsky MP, Xie C, Dewberry LC, Sitzman TJ. Body contouring in adolescents after bariatric surgery. Surg Obes Relat Dis. 2020 Jan;16(1):137-142. doi: 10.1016/j.soard.2019.09.063. Epub 2019 Sep 18. PMID 31668945
- [Background] Aldaqal SM, Samargandi OA, El-Deek BS, Awan BA, Ashy AA, Kensarah AA. Prevalence and desire for body contouring surgery in postbariatric patients in saudi arabia. N Am J Med Sci. 2012 Feb;4(2):94-8. doi: 10.4103/1947-2714.93386. PMID 22408756
- [Background] Hult M, Bonn SE, Brandt L, Wiren M, Lagerros YT. Women's Satisfaction with and Reasons to Seek Bariatric Surgery-a Prospective Study in Sweden with 1-Year Follow-up. Obes Surg. 2019 Jul;29(7):2059-2070. doi: 10.1007/s11695-019-03834-3. PMID 30955156